CLINICAL TRIAL: NCT02068261
Title: Computerized Working Memory Training in Adults With Substance Abuse and Executive Function Deficits: A Randomised Controlled Trial.
Brief Title: Working Memory Training in Adults With Substance Abuse and Executive Function Deficits.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro Läns Landsting (Other Government)
Responsible Party: Principal Investigator, Rickard Ahlberg, Clinical psychologist, doctoral student., Örebro Läns Landsting
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA02
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Substance Abuse; Executive Dysfunction; Anxiety; Depression; Antisocial Personality; Reading Disabilities
MeSH Terms: conditions — Substance-Related Disorders; Anxiety Disorders; Depression; Antisocial Personality Disorder; Dyslexia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed working memory training (Experimental): 30-40 minutes of Cogmed computerized working memory training 3-5 days a week for 5-8 weeks. Every training session consists of a set of visual- and verbal working memory tasks that are trained on during the session.
  Interventions: Behavioral: Computerized Cogmed working memory training
- Treatment as usual (Active Comparator): Treatment as usual can consist of medication, psychotherapy, counseling, and psychological assessment. After a 8 week period participants in this arm well be offered Cogmed working memory training.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Computerized Cogmed working memory training — Computerized working memory training with Cogmed QM software. The QM software consists of a set of verbal and visual working memory tasks which is trained for 25-40 minutes each session.
  Arms: Cogmed working memory training
Behavioral: Treatment as usual — Treatment as usual can consist of medication, psychotherapy, counseling, and psychological assessment.
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to evaluate the effects of a computerized working memory training program on substance abuse, psychosocial functioning, cognitive performance and psychiatric problems in adults with substance abuse and attention problems.

DETAILED DESCRIPTION:
The primary aim of this study is to examine the effects of 5 weeks of computerized working memory training on substance abuse. Secondary aims are to explore whether effects are mediated by changes in executive functions and/or moderated by personality. Also, effects on measures of psychosocial functioning, depression, anxiety and attention will be explored. Follow-up assessment will be conducted at 6 months post training.

ELIGIBILITY:
Inclusion Criteria:

* Treatment seeking adults with substance abuse and executive function deficits.

Exclusion Criteria:

* Acute intoxication or abstinence symptoms of any substance.
* Psychosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in substance abuse measured with Substance abuse scales in Adult Self Report (ASR; ASEBA). | Baseline and at 25 weeks

SECONDARY OUTCOMES:
Change from baseline in Adult Self Report (ASR; ASEBA) Attention problems scale. | Baseline and at 25 weeks
Change from baseline in Adult Self Report (ASR; ASEBA) Internalizing index. | Baseline and at 25 weeks
Change from baseline in Adult Self Report (ASR; ASEBA) Externalizing index. | Baseline and at 25 weeks
Change from baseline in Adult Self Report (ASR; ASEBA) Adaptive functioning scales. | Baseline and at 25 weeks
Change from baseline in Executive functioning measured with Behavior Rating Inventory of Executive Function-Adult (BRIEF-A). | Baseline and at 25 weeks
Change from baseline in verbal working memory measured with performance on Digit span. | Baseline and at 25 weeks
Change from baseline in visual working memory measured with performance on Span board. | Baseline and at 25 weeks
Change from baseline in focused attention measured with performance on Conners Continuous Performance Test-II (CCPT-II). | Baseline and at 25 weeks
Change from baseline in vigilance measured with performance on Conners Continuous Performance Test-II (CCPT-II). | Baseline and at 25 weeks
Change from baseline in reading speed measured with performance on Reading speed in Diagnostic Reading and Writing Test (DLS; Swedish version). | Baseline and at 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Kjellin, Docent, Study Director — Örebro Läns Landsting
Locations (1):
- Psychiatric Research Centre, Örebro, Örebro County, Sweden